CLINICAL TRIAL: NCT02150694
Title: Local Haemodynamic Effects of Apelin Agonists and Antagonists in Man in Vivo
Acronym: HEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Aimee Brame MRCP, Research Fellow, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HEAP Study
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Apelin agonist infusion (Experimental): Studies to measure change in blood flow in response to apelin agonists (1/10/100nmol) using forearm venous occlusion plethysmography and Aellig hand vein technique.
  Interventions: Procedure: Forearm venous occlusion plethysmography; Procedure: Aellig hand vein technique; Other: Apelin agonist infusion
- Apelin receptor antagonist infusion (Experimental): Aellig hand vein technique will be used to investigate the change in vein diameter in response to an apelin blocking agent
  Interventions: Procedure: Aellig hand vein technique; Other: Apelin receptor antagonist infusion
- Apelin agonist/antagonist co-infusion (Experimental): Forearm blood flow study to measure blood flow by forearm venous occlusion plethysmography following intraarterial infusion of apelin receptor agonists and antagonist.
  Interventions: Procedure: Forearm venous occlusion plethysmography; Other: Apelin agonist infusion; Other: Apelin receptor antagonist infusion

INTERVENTIONS:
Procedure: Forearm venous occlusion plethysmography — Forearm venous occlusion plethysmography to study to measure forearm blood flow during intra-arterial infusion of the apelin peptides.
  Arms: Apelin agonist infusion; Apelin agonist/antagonist co-infusion
Procedure: Aellig hand vein technique — Hand vein measurements will be used to assess the response to apelin peptides and apelin receptor blocker in the human hand vein vascular bed.
  Arms: Apelin agonist infusion; Apelin receptor antagonist infusion
Other: Apelin agonist infusion — Escalating doses of apelin (1/10/100nmol/min) will be administered.
  Arms: Apelin agonist infusion; Apelin agonist/antagonist co-infusion
Other: Apelin receptor antagonist infusion — Dose finding study (range 1-300nmol/min) and co-infusion study with apelin peptides
  Arms: Apelin agonist/antagonist co-infusion; Apelin receptor antagonist infusion

SUMMARY:
Apelins are substances which occur naturally in the body, and have an important role in heart disease. They have been shown to make blood vessels dilate, and improve the way the heart works.

The investigators have devised 2 sets of experiments to investigate how the apelins affect blood vessels.

In the first group of experiments,the investigators will give healthy volunteers up to 3 different apelin substances, and use special research techniques to see how they affect the way that blood vessels work in the forearm.

In the second group of experiments, the apelins will be given along with another form of apelin which blocks the effects of apelin in laboratory experiments. The investigators want to see if it blocks the effects of apelin in healthy humans.

The investigators intend to test the hypothesis that:

Apelin agonists are vasodilators in human resistance vessels, this effect will be blocked by an apelin receptor antagonist.

This study will help us to understand more about how apelins work, and to suggest how they might be used to treat heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years
* Non-regular smoking (<5 cigarettes per week)
* If female, postmenopausal or on days 2-9 of menstrual cycle

Exclusion Criteria:

* Hypertension (sustained BP >160/100mmHg)
* Ischaemic Heart Disease
* Renal, respiratory or neurological disease
* Diabetes mellitus
* BMI >30, BMI <18
* Pregnant
* Smoker
* Use of vasoactive medication or NSAIDS/aspirin within 48 hours of study.
* Current involvement in other research studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by forearm plethysmography in response to infused vasodilators | 2-3 hours
Change in hand vein diameter measured by Aellig hand vein technique, in response to study peptides | 2-3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ian B Wilkinson, FRCP DM, Study Director — University of Cambridge; Anthony P Davenport, MA PhD, Study Director — University of Cambridge
Locations (1):
- Vascular Research Unit, Cambridge, United Kingdom